CLINICAL TRIAL: NCT05167838
Title: A Comparative Study Between Fresh and Frozen Embryo Transfer in Cases of Polycystic Ovaries Syndrome (PCOS) Patients Undergoing in Vitro Fertilization (IVF) Treatment for Infertility as Regards Clinical Pregnancy Rate and IVF Outcome
Brief Title: Comparative Study Between Fresh and Frozen Embryo Transfer in PCOS Patients Undergoing IVF Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Mahmoud Eid, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cairo University obgyn
Record Dates: First submitted 2021-11-23; First posted 2021-12-22 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: IVF
Keywords: IVF-Fresh ET-FET-clinical pregnancy

STUDY DESIGN:
Intervention Model Description: Group 1; Fresh embryo transfer in PCO patients Group 2: Frozen ET in PCO patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Fresh embryo transfer group
  Interventions: Procedure: fresh embryo transfer
- Group B (Experimental): Frozen embryo transfer group
  Interventions: Procedure: Frozen embryo transfer

INTERVENTIONS:
Procedure: fresh embryo transfer — 55 patients undergoing fresh embryo transfer after ovarian stimulation followed by luteal phase support
  Arms: group A
Procedure: Frozen embryo transfer — 55 patients undergoing frozen embryo transfer after ovarian stimulation followed by cryopreservation of all embryos and transfer in another cycle.
  Arms: Group B

SUMMARY:
The objective of our study is to compare in vitro fertilization (IVF) outcomes between fresh embryo transfer (ET) and frozen-thawed ET in women with polycystic ovary syndrome (PCOS).

DETAILED DESCRIPTION:
Eligible women will be randomized to two groups in a ratio of 1:1 . Both the patients and the clinicians will be aware of the allocated arm. The patients (110) will be equally randomized into two groups:

Group A will undergo a day 3 fresh embryo transfer after ovarian stimulation, luteal phase support will be started just after follicular aspiration. Group B will have all of their embryo cryopreserved after ovarian stimulation with no luteal phase support after the aspiration and then undergo a frozen-thawed day 3 embryo transfer.

Controlled ovarian stimulation will be done using the gonadotropin releasing hormone (GnRH) antagonist protocol then human chorionic gonadotropin( HCG) 5000 IU trigger for final oocyte maturation.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with PCOS according to modified Rotterdam criteria which includes menstrual abnormalities combined with either hyperandrogenism (hirsutism diagnosed by modified Ferriman-Gallwey score or elevated total testosterone level) or polycystic ovaries.
* Women ages ≥20 and <40years old.
* BMI less than 35.
* Women who have a history of infertility.
* All patients will receive adjuvant drugs for ovulation induction (metformin from preceding cycle, cabergoline 1 tab daily for 8 days and 500 cc colloid solution on day of ovum pick up).

Exclusion Criteria:

* History of unilateral oophorectomy.
* Uterine abnormalities such as a malformed uterus (unicornuate, septate uterus), adenomyosis, submucous myoma or intrauterine adhesion.
* Severe male factor for infertility such as azoospermia.
* History of repeated ICSI trials failure.
* Women who are unable to comply with the study procedures.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 35 days after embryo transfer
  Transvaginal Ultrasound to detect gestational sac(GS)

SECONDARY OUTCOMES:
Chemical pregnancy rate | 14 days after embryo transfer.
  Serum β-human chorionic gonadotropin (HCG) will be measured to determine pregnancy after embryo transfer.
Early ovarian hyperstimulation syndrome rate(OHSS rate) | 3 days after follicular aspiration
  Abdominal ultrasound ,Hematocrit
Ectopic pregnancy rate | 14 days for BHCG , vaginal US 3 weeks after transfer
  BHCG then doubling after 48 hours ,vaginal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Mo Eid, MD, Principal Investigator — Cairo U
Locations (1):
- Marwa Eid, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided